CLINICAL TRIAL: NCT02604160
Title: A Multiple-Dose, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of LY3113593 in Patients Receiving Hemodialysis
Brief Title: A Study of LY3113593 in Participants With Chronic Kidney Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16045; I7C-MC-FEAC (Other: Eli Lilly and Company)
Record Dates: First submitted 2015-11-11; First posted 2015-11-13 (Estimated); Results first posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-08

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant
Masking Description: single-blind participant only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- LY3113593 (Experimental): Escalating doses of LY3113593 administered by intravenous (IV) infusion once every 4 weeks (Q4W) on (Day 1 and 29) in part A.
  Interventions: Drug: LY3113593
- Placebo (Placebo Comparator): 0.9% saline, administered by intravenous (IV) infusion once Q4W (Day 1 and 29) in part A.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3113593 — Administered by slow intravenous (IV) infusion.
  Arms: LY3113593
Drug: Placebo — Administered by slow intravenous (IV) infusion.
  Arms: Placebo

SUMMARY:
This study is not intended to treat anemia of chronic kidney disease but to determine the safety of the study drug, LY3113593.

The study will also evaluate how much of the study drug gets into the blood stream, how long it takes the body to remove the study drug, and what effect the study drug has on the body.

The study consists of up to three parts. Participants may only enroll in one part. Participants will receive up to four injections of LY3113593 or placebo into a vein. The study will last up to about 26 weeks including screening and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Receiving hemodialysis regularly (at least 3 times per week) for at least 4 months
* Have a hemoglobin value (taken prior to dialysis, if taken on a dialysis day) greater than or equal to 9.5 grams per deciliter (g/dL) and less than or equal to 11.0 g/dL at screening
* Have been receiving erythropoiesis stimulating agent (ESA) injections for at least 4 weeks and are willing to stop the injections for approximately 8 weeks

Exclusion Criteria:

* Have another health condition that may put the participant at risk or that the study doctor feels would make the participant unsuitable for the study
* Currently taking part in another study
* Have recently (within 30 days) completed a study or have previously taken part in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-11-17; Primary Completion 2016-06-22 (Actual); Study Completion 2016-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (5):
- United States (5):
  - Orlando Clinical Research Center, Orlando, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Northwest Louisiana Nephrology, Shreveport, Louisiana
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Clinical Advancement Center, PLLC, San Antonio, Texas

REFERENCES:
- [Derived] Sheetz M, Barrington P, Callies S, Berg PH, McColm J, Marbury T, Decker B, Dyas GL, Truhlar SME, Benschop R, Leung D, Berg J, Witcher DR. Targeting the hepcidin-ferroportin pathway in anaemia of chronic kidney disease. Br J Clin Pharmacol. 2019 May;85(5):935-948. doi: 10.1111/bcp.13877. Epub 2019 Mar 4. PMID 30677788
- See also: Click here for more information about this study: A Study of LY3113593 in Participants With Chronic Kidney Disease — http://www.lillytrialguide.com/EN/studies/kidney-disease/feac

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Part A of the study, a dose stopping criterion was met leading to early conclusion of the study.
Groups:
- Placebo: 0.9% saline, administered by intravenous (IV) infusion once every four weeks (Q4W) (Day 1 and 29) in part A.
- LY3113593: 50 milligram (mg) of LY3113593 administered by IV infusion Q4W (Day 1 and 29) in part A.
Period: Overall Study
Arm/Group | Placebo | LY3113593
Started | 2 | 5
Received at Least One Dose of Study Drug | 2 | 5
Completed | 2 | 3
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | LY3113593 | Total
Number analyzed (Participants) | 2 | 5 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 2 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 1 | 3 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 0 | 3 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration
Description: A summary of other non-serious adverse events (AEs) and all serious adverse events, regardless of causality, is located in the reported adverse events section.
Time Frame: Baseline through Day 29
Population: All participants who received at least one dose of study drug or placebo, and have at least one post dose safety assessment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: 0.9% saline of placebo administered by IV infusion Q4W (Day 1 and 29) in part A.
- LY3113593: 50 mg of LY3113593 administered by IV infusion Q4W (Day 1 and 29) in part A.
Arm/Group | Placebo | LY3113593
Number analyzed (Participants) | 2 | 5
Participants | 0 | 1

2. Secondary Outcome: Pharmacokinetics (PK): Maximum Drug Concentration (Cmax) of LY3113593
Time Frame: Predose; 0.5, 4 hours post-dose
Population: All participants who received at least one dose of study drug and have evaluable PK data. PK was not assessed in placebo.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | LY3113593
Number analyzed (Participants) | 5
nanogram/milliliter (ng/mL)
  Day 1 | 11934 (30)
  Day 29 | 13567 (42)

3. Secondary Outcome: PK: Area Under the Concentration Versus Time (AUCτ)
Description: Area under the concentration versus time (AUCτ) is the AUC over the dosing interval (Q4W)
Time Frame: Predose; 0.5, 4 hours post-dose
Population: All participants who received at least one dose of study drug and had evaluable PK data. PK was not assessed in placebo.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram.hour/milliliter (ug*h/mL)
Groups:
- LY3113593: 50 mg of LY3113593 administered by IV infusion Q4W on (Day 1 and 29) in part A.
Arm/Group | LY3113593
Number analyzed (Participants) | 5
microgram.hour/milliliter (ug*h/mL)
  Day 1 | 2281 (36)
  Day 29 | 2707 (36)

4. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline to Week 8 in Hemoglobin (Hb)
Time Frame: Predose; 0.5, 4 hours post-dose
Population: Zero participants were analyzed; data not collected. Change from baseline to week 8 in Hemoglobin (Hb) was not assessed since study was concluded early at part A.
Arm/Group | Placebo | LY3113593
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Anti-LY3113593 Antibodies Detection
Description: Participants with a detection of anti-LY3113593 antibodies at baseline and post-baseline time point at the following levels of 1:20, 1:40 or 1:80 titer.
Time Frame: Day 1: Predose; Day 15, 29, 57, 85 and 113
Population: All participants who received at least one dose of study drug, and have at least one post dose safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | LY3113593
Number analyzed (Participants) | 2 | 5
Participants
  Day 1 Predose; 1:80 Titer | 1 | 0
  Day 15 ± 2 days; 1:20 Titer | 1 | 0
  Day 29 ± 2 days; 1:80 Titer | 1 | 0
  Day 57 ± 2 days; 1:40 Titer | 1 | 0
  Day 85 ± 2 days; 1:40 Titer | 1 | 0
  Day 113; ± 2 days; 1:40 Titer | 0 | 0

ADVERSE EVENTS:
Groups:
- Placebo: 0.9% saline, administered by slow IV infusion Q4W (Day 1 and 29) in part A.
- LY3113593: 50 mg of LY3113593 administered by slow IV infusion Q4W (Day 1 and 29) in part A.
Arm/Group | Placebo | LY3113593
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/5
Other Adverse Events (participants affected / at risk) | 2/2 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | LY3113593 (N=5)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=2) | LY3113593 (N=5)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Hyperparathyroidism secondary (Endocrine disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
In Part A of the study, a dose stopping criterion was met leading to early conclusion of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days